CLINICAL TRIAL: NCT04370561
Title: a Prospective Randomized Study on the Outcome Following Osteosynthesis of Distal Fibula Fracture Using Semitubular Plate in AO Technique vs. Polyaxial Locking Plates
Brief Title: Outcome Following Semitubular Plate vs. Polyaxial Locking Plates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Principal Investigator, Dr. Chlodwig Kirchhoff, Clinical Professor, Technical University of Munich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ActiveAnkle_0815
Record Dates: First submitted 2020-04-20; First posted 2020-05-01 (Actual); Last update posted 2020-05-05 (Actual); Status verified 2020-05

CONDITIONS: Ankle Fractures
MeSH Terms: conditions — Ankle Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1/3 tubular plate (Active Comparator): Standard care according to AO guidelines using the Implant "1/3 tubular plate"
  Interventions: Procedure: ORIF non-locking
- Active ankle plate (Active Comparator): Actual care using the new implant using the Implant "Active ankle plate"
  Interventions: Procedure: ORIF locking

INTERVENTIONS:
Procedure: ORIF non-locking — Open reduction and internal fixation using 1/3 tubular plate
  Arms: 1/3 tubular plate
Procedure: ORIF locking — Open reduction and internal fixation using active ankle polyaxial locking plate
  Arms: Active ankle plate

SUMMARY:
In this prospective study, all patients with distal fibula fractures (AO 44 B1.1, B1.2, B1.3), with indication for surgery were included. Patients were randomized to either the DePuy Synthes® one-third semitubular plate (Group I) or NEWCLIP TECHNICS, Active Ankle® polyaxial locking plate (Group II). In Group II early weight bearing was allowed after two weeks postoperatively. Primary outcome parameter was function of the ankle joint, assessed by the Olerud and Molander ankle score (OMAS), Foot and Ankle outcome score (FAOS) and Karlsson and Peterson Scoring System for Ankle function (KPSS). Secondary outcome parameter were postoperative complications. Superficial wound infection, delayed wound healing, mechanically prominent implant, skin irritations were considered as minor and deep wound infection, material loosening, loss of reduction were regarded as major complications requiring revision surgery. Clinical and radiological follow-up were performed 6 and 12 weeks, 6 months and 1 year postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 65 years
* Fracture of the distal fibula (AO 44 B1.1, B1.2, B1.3)
* Written informed consent

Exclusion Criteria:

* Pregnancy
* mental disorders
* comprehensive legal support.
* pathological and/or osteoporotic fracture
* open fracture

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Ankle function | 12 month
  Clinical objective ankle function assessed by Olerud and Molander ankle score (OMAS)

SECONDARY OUTCOMES:
Ankle function | 12 month
  Clinical objective ankle function assessed by Foot and Ankle outcome score (FAOS)

CONTACTS AND LOCATIONS:
Overall Officials: Chlodwig Kirchhoff, MD, Principal Investigator — Klinik für Unfallchirurgie, Klinikum rechts der Isar, TU München

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zyskowski M, Wurm M, Greve F, Pesch S, von Matthey F, Pfluger P, Cronlein M, Biberthaler P, Kirchhoff C. Is early full weight bearing safe following locking plate ORIF of distal fibula fractures? BMC Musculoskelet Disord. 2021 Feb 9;22(1):159. doi: 10.1186/s12891-021-04009-x. PMID 33563235